CLINICAL TRIAL: NCT01081275
Title: Rehabilitating Extremity Use After Multiple Sclerosis
Brief Title: Improving Hand Use in Multiple Sclerosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Victor W. Mark, Associate Professor, National Multiple Sclerosis Society
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RG 4221-A-2
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; MS; CI Therapy; CIMT; Constraint-Induced Movement Therapy; Complementary and Alternative Medicine; CAM; Physical Therapy; Occupational Therapy; Relaxation; Exercise; Massage; Yoga; Pool Therapy; Aquatherapy; Aquatic Therapy
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity | interventions — Constraint Induced Movement Therapy; Complementary Therapies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CI Therapy (Active Comparator): CI therapy involves repetitive practice with the more-affected hand on typical daily living activities (such as stacking objects, pouring, moving objects) for 3.5 hours per day, along with physical restraint of the better hand to keep it from assisting, and home practice exercises.
  Interventions: Behavioral: CI Therapy
- CAM treatments (Active Comparator): CAM treatments are holistic physical treatments designed to work on the entire body to improve quality of life and overall health. This study will use yoga, relaxation exercises, aquatherapy (pool therapy), and massage.
  Interventions: Behavioral: CAM treatments

INTERVENTIONS:
Behavioral: CI Therapy — CI Therapy will be given for 3.5 hours per day, Monday-Friday, for 2 consecutive weeks.
  Other Names: Constraint-Induced Movement therapy
  Arms: CI Therapy
Behavioral: CAM treatments — CAM treatments will be given for 3.5 hours per day, Monday-Friday, for 2 consecutive weeks.
  Other Names: Complementary and Alternative Medicine
  Arms: CAM treatments

SUMMARY:
This study will compare two different kinds of physical therapy to improve use of the hands in individuals with multiple sclerosis (MS). One treatment will be Constraint-Induced Movement therapy (CI therapy), the other will be a set of Complementary and Alternative Medicine (CAM) treatments (yoga, relaxation exercises, aquatherapy, massage). The study will determine which of the two forms of treatment is more successful for improving hand use.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) frequently causes reduced use of one of the hands, and as a result, much of daily living activities are conducted only by the other hand, leaving the person effective one-handed. Nonetheless, reduced hand use can be improved for extended amounts of time with specific forms of physical therapy, as long as persons with MS have the ability to perform the training tasks.

This study will randomize persons with MS who have relatively reduced use of one of the hands to either CI therapy or CAM treatments. Treatment in either program will be for 2 consecutive weeks, 3.5 hours per day (Monday-Friday), under the direct supervision of a specially trained therapist. Before starting, participants will also undergo comprehensive medical and physical exam screening and brain MRI scan. The same evaluations will be performed after treatment to learn whether any of these have changed as a result of treatment.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of non-relapsing multiple sclerosis (primary progressive MS, secondary progressive MS)
* reduced use of one of the hands because of MS
* ability to pick up and release a small object with the more-affected hand when requested
* can travel to the treatment program at the University of Alabama at Birmingham (UAB)
* can undergo treatment for 2 weeks (Monday-Friday), 3.5 hours per day
* can undergo MRI scan
* any kind of medication used for MS is allowed except spasticity medicine

Exclusion Criteria:

* disease relapse in the past 3 months
* pregnancy
* marked pain with arm movement
* severe uncontrolled medical illness
* simultaneous treatment with another form of physical therapy

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2010-02; Primary Completion 2016-02 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Motor Activity Log (MAL) | Before treatment, and immediately, 6 months, and 12 months after the end of treatment.
  The MAL is a structured interview on the amount and quality of the more-affected hand use during daily living activities.

SECONDARY OUTCOMES:
Wolf Motor Function Test (WMFT) | Before treatment, and immediately, 6 months, and 12 months after the end of treatment.
  The WMFT evaluates how fast the more-affected hand can complete several activities that resemble those in the home (such as bringing a can to the lips).
MSFC (Multiple Sclerosis Composite Measure) | Before treatment, and immediately, 6 months, and 12 months after the end of treatment.
  The MSFC evaluates memory, hand dexterity, and walking (for individuals who can walk without another person's assistance).
SARA (Scale for the Assessment and Rating of Ataxia) | Before treatment, and immediately, 6 months, and 12 months after the end of treatment.
  The SARA evaluates the control of ataxia (incoordination, tremor) of hand movements.
EDSS (Expanded Disability Status Scale) | Before treatment, and immediately, 6 months, and 12 months after the end of treatment.
  The EDSS is the world-wide standard to evaluate physical capability in persons with MS.
Fatigue Severity Scale (FSS) | Before treatment, and immediately, 6 months, and 12 months after the end of treatment.
  The FSS evaluates the degree of overall fatigue experienced by the person with MS.
MSIS-29 (Multiple Sclerosis Impact Scale) | Before treatment, and immediately, 6 months, and 12 months after the end of treatment.
  The MSIS-29 is a questionnaire that evaluates the impact of MS on daily living activities and quality of life.
MSSS-88 (Multiple Sclerosis Spasticity Scale) | Before treatment, and immediately, 6 months, and 12 months after the end of treatment.
  The MSSS-88 examines the extent of stiffness (spasticity) of the arm in persons with MS.
Baecke Activity Questionnaire | Before treatment, and immediately, 6 months, and 12 months after the end of treatment.
  The Baecke evaluates the impact of disease upon employment and leisure time activities.

CONTACTS AND LOCATIONS:
Overall Officials: Victor W Mark, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Background] Mark VW, Taub E, Bashir K, Uswatte G, Delgado A, Bowman MH, Bryson CC, McKay S, Cutter GR. Constraint-Induced Movement therapy can improve hemiparetic progressive multiple sclerosis. Preliminary findings. Mult Scler. 2008 Aug;14(7):992-4. doi: 10.1177/1352458508090223. Epub 2008 Jun 23. PMID 18573826
- [Derived] Barghi A, Allendorfer JB, Taub E, Womble B, Hicks JM, Uswatte G, Szaflarski JP, Mark VW. Phase II Randomized Controlled Trial of Constraint-Induced Movement Therapy in Multiple Sclerosis. Part 2: Effect on White Matter Integrity. Neurorehabil Neural Repair. 2018 Mar;32(3):233-241. doi: 10.1177/1545968317753073. PMID 29668401
- [Derived] Mark VW, Taub E, Uswatte G, Morris DM, Cutter GR, Adams TL, Bowman MH, McKay S. Phase II Randomized Controlled Trial of Constraint-Induced Movement Therapy in Multiple Sclerosis. Part 1: Effects on Real-World Function. Neurorehabil Neural Repair. 2018 Mar;32(3):223-232. doi: 10.1177/1545968318761050. PMID 29668399